CLINICAL TRIAL: NCT04126343
Title: A Single-Center, Randomized, Placebo-Controlled, 3 Treatment Period Crossover Study to Assess the Effect of Padsevonil on Cardiac Repolarization (QTc Interval) (Using Moxifloxacin as a Positive Control) in Healthy Study Participants
Brief Title: A Study to Test the Cardiac Effects of Padsevonil in Healthy Study Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on available data, UCB has decided to stop development of padsevonil as adjunctive treatment of focal-onset seizures
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0050; 2019-002797-31 (EudraCT Number)
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Healthy Study Participants
Keywords: Healthy study participants; Padsevonil; Moxifloxacin; Cardiac repolarization
MeSH Terms: interventions — padsevonil; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Padsevonil (Experimental): Study participants randomized to this arm will receive assigned doses of padsevonil twice daily. On Day 8 padsevonil will be administered in the morning, and placebo will administered in the evening.
  Interventions: Drug: Padsevonil; Drug: Placebo
- Placebo (Placebo Comparator): Study participants randomized to this arm will receive placebo twice daily to maintain the blinding.
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Study participants randomized to this arm will receive padsevonil-placebo twice daily. On Day 8 placebo will be administered in the morning, and moxifloxacin will administered in the evening.
  Interventions: Drug: Moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: Padsevonil — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  * Study participants will receive padsevonil in a pre-specified dosing sequence during the Treatment Period
  Arms: Padsevonil
Drug: Moxifloxacin — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  * Study participants will receive moxifloxacin once during the Treatment Period
  Arms: Moxifloxacin
Drug: Placebo — * Pharmaceutical form: Film-coated tablet
  * Route of administration: Oral use
  * Study participants will receive placebo in a pre-specified sequence during the Treatment Period to match padsevonil and maintain the blinding

SUMMARY:
The purpose of the study is to evaluate the effects on cardiac repolarization of high-dose padsevonil (PSL) in comparison to placebo in healthy study participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent form (ICF)
* Participant who is overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Body weight of at least 50 kilogram (kg) (males) or 45 kg (females) and body mass index (BMI) within the range 18 to 30 kg/m2 (inclusive)
* Male and/or female:

A male study participant must agree to use contraception during the Treatment Period and for at least 90 days after the last dose of study medication and refrain from donating sperm during this period

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the Treatment Period and for at least 90 days after the last dose of study medication

Exclusion Criteria:

* Participant has a known hypersensitivity to any components of the study medication or comparative drugs as stated in this protocol or history of tendon pathology secondary to use of quinolone antibiotics
* Participant has a history of unexplained syncope or a family history of sudden death due to long QT syndrome
* Participant has a present condition of respiratory or cardiovascular disorders, eg, cardiac insufficiency, coronary heart disease, hypertension, arrhythmia, tachyarrhythmia, or myocardial infarction
* Past or intended use of over-the-counter (OTC) or prescription medication including herbal medications within 2 weeks or 5 half-lives prior to dosing.
* Participant has used hepatic enzyme-inducing drugs (eg, glucocorticoids, phenobarbital, isoniazid, phenytoin, rifampicin, etc) within 2 months prior to the first dose of study medication
* Participant has previously received padsevonil (PSL) in this or any other study
* Participant has any clinically relevant electrocardiogram (ECG) finding at the Screening Visit or at Baseline. Participant has an abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risks associated with participating in the study. In addition, any participant with any of the following findings will be excluded:

  1. QT interval corrected for heart rate using the Fridericia method (QTcF) ≥450 ms (on mean of triplicate ECG recordings);
  2. Other conduction abnormalities (defined as PR interval >220 ms);
  3. QRS interval >109 ms;
  4. Any rhythm other than sinus rhythm;
  5. Any history of Wolff-Parkinson-White Syndrome, Brugada Syndrome, unexplained syncope, or ventricular tachycardia;
  6. Family history of QTc prolongation or of unexplainable sudden death at <50 years of age
* Participant has made a blood or plasma donation or has had a comparable blood loss (>450 mL) within 30 days prior to the Screening Visit. Blood donation during the study is not permitted

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0050 001, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in October 2019 and concluded in May 2020.
Pre-assignment Details: The Participant Flow refers to the Safety Set.
Groups:
- Treatment Sequence: ABC: Padsevonil (PSL) Treatment Period (Treatment A)- participants received PSL 100 milligrams (mg) to 400 mg, orally twice daily (bid) during the 11 Days PSL Treatment Period. On Day 8, the Target Dose Day, participants received PSL 400 mg in the morning only and placebo in the afternoon.
  Placebo Treatment Period (Treatment B)-participants received Placebo matched to PSL Treatment Period doses, bid up to Day 11.
  Moxifloxacin (MXF) Treatment Period (Treatment C)- participants received placebo matched to PSL Treatment Period doses, bid up to Day 11. On Day 8, the Target Dose Day, participants received MXF 400 mg in the morning and placebo in the afternoon.
  Participants received PSL, Placebo, and MXF treatments at the first, the second and the third treatment periods respectively, with a minimum 7-day washout period between each treatment periods.
- Treatment Sequence: ACB: Participants received PSL, MXF, and Placebo treatments at the first, the second and the third treatment periods respectively, with a minimum 7-day washout period between each treatment periods.
- Treatment Sequence: BAC: Participants received Placebo, PSL, and MXF treatments at the first, the second and the third treatment periods respectively, with a minimum 7-day washout period between each treatment periods.
- Treatment Sequence: BCA: Participants received Placebo, MXF, and PSL treatments at the first, the second and the third treatment periods respectively, with a minimum 7-day washout period between each treatment periods.
- Treatment Sequence: CAB: Participants received MXF, PSL, and Placebo treatments at the first, the second and the third treatment periods respectively, with a minimum 7-day washout period between each treatment periods.
- Treatment Sequence: CBA: Participants received MXF, Placebo, and PSL treatments at the first, the second and the third treatment periods respectively, with a minimum 7-day washout period between each treatment periods.
Period: Overall Study
Arm/Group | Treatment Sequence: ABC | Treatment Sequence: ACB | Treatment Sequence: BAC | Treatment Sequence: BCA | Treatment Sequence: CAB | Treatment Sequence: CBA
Started | 9 | 9 | 9 | 9 | 9 | 9
Completed Padsevonil Period | 9 | 9 | 9 | 7 | 9 | 8
Completed Placebo Period | 9 | 7 | 9 | 9 | 7 | 9
Completed Moxifloxacin Period | 8 | 9 | 7 | 9 | 9 | 9
Completed | 6 | 5 | 6 | 5 | 6 | 5
Not Completed | 3 | 4 | 3 | 4 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Related to COVID-19 pandemic | 3 | 4 | 3 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all study participants who received at least 1 dose of study medication.
Groups:
- Treatment Sequence: ABC: Padsevonil (PSL) Treatment Period (Treatment A) participants received PSL 100 milligrams (mg) to 400 mg, orally twice daily (bid) during the 11 Days PSL Treatment Period. On Day 8, the Target Dose Day, participants received PSL 400 mg in the morning only and placebo in the afternoon.
  Placebo Treatment Period (Treatment B) participants received Placebo matched to PSL Treatment Period doses, bid up to Day 11.
  Moxifloxacin (MXF) Treatment Period (Treatment C) participants received placebo matched to PSL Treatment Period doses, bid up to Day 11. On Day 8, the Target Dose Day, participants received MXF 400 mg in the morning and placebo in the afternoon.
  Participants received PSL, Placebo, and MXF treatments at the first, the second and the third treatment periods respectively, with a minimum 7-day washout period between each treatment periods.
Arm/Group | Treatment Sequence: ABC | Treatment Sequence: ACB | Treatment Sequence: BAC | Treatment Sequence: BCA | Treatment Sequence: CAB | Treatment Sequence: CBA | Total Title
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 9 | 8 | 9 | 9 | 9 | 9 | 53
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (6.9) | 30.2 (9.5) | 38.4 (7.1) | 37.0 (7.6) | 36.8 (9.9) | 32.4 (5.6) | 35.1 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 1 | 0 | 3
  Male | 8 | 8 | 9 | 9 | 8 | 9 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 0 | 0 | 0 | 1 | 3
  Black or African American | 1 | 0 | 0 | 2 | 0 | 0 | 3
  White | 7 | 7 | 9 | 7 | 8 | 5 | 43
  Other/mixed | 0 | 1 | 0 | 0 | 1 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Placebo-corrected Change From Baseline in QTcF on Day 8 for Padsevonil
Description: Placebo-corrected change from Baseline in corrected QT interval (QTc), based on Fridericia's correction (QTcF) method (ΔΔQTcF) evaluated during the Target Dose Day of the padsevonil and placebo Treatment Periods, using linear mixed-effects model analysis.
Time Frame: Day 8 : 0.75, 0.5, 0.25 hours predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24 hours postdose
Population: The QT/QTc Set included all study participants in the SS with measurements at Baseline as well as on-treatment with at least 1 postdose time point with a valid change-from Baseline QTcF (ΔQTcF) value. Here, number of participants were included who were evaluable for the assessment.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds (ms)
Groups:
- Padsevonil (QT/QTc Set): Participants received PSL 100 mg to 400 mg orally bid during the 11 Days PSL Treatment Period. On Day 8, the Target Dose Day, participants received PSL 400 mg in the morning only and placebo in the afternoon. Participants formed the QT/corrected QT interval (QTc) Set.
Arm/Group | Padsevonil (QT/QTc Set)
Number analyzed (Participants) | 46
milliseconds (ms)
  0.75 hour Predose | -1.2 [-4.0 to 1.6]
  0.5 hour Predose | -1.8 [-4.7 to 1.1]
  0.25 hour Predose | -0.7 [-3.5 to 2.1]
  0.25 hour Postdose | -0.5 [-3.6 to 2.6]
  0.5 hour Postdose | -0.9 [-3.8 to 1.9]
  1 hour Postdose | -1.8 [-4.6 to 1.0]
  1.5 hours Postdose | -1.3 [-4.2 to 1.5]
  2 hours Postdose | -1.8 [-4.7 to 1.2]
  3 hours Postdose | -2.5 [-6.0 to 1.0]
  4 hours Postdose | -1.5 [-4.6 to 1.6]
  6 hours Postdose | -0.6 [-3.8 to 2.5]
  8 hours Postdose | -2.0 [-5.3 to 1.3]
  12 hours Postdose | -2.9 [-7.1 to 1.2]
  18 hours Postdose | -4.9 [-8.1 to -1.7]
  24 hours Postdose | -1.5 [-4.8 to 1.8]

2. Secondary Outcome: Placebo-corrected Change From Baseline in QTcF After a Single Dose of Moxifloxacin on Day 8
Description: Placebo-corrected change from Baseline in corrected QT interval (QTc), based on Fridericia's correction (QTcF) method (ΔΔQTcF) evaluated during the Target Dose Day of the moxifloxacin and placebo Treatment Periods, using linear mixed-effects model analysis.
Time Frame: Day 8 : 0.75, 0.5, 0.25 hours predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- Moxifloxacin (QT/QTc Set): Participants received placebo matched to PSL Treatment Period doses, bid up to Day 11.
  On Day 8, the Target Dose Day, participants received MXF 400 mg in the morning and placebo in the afternoon. Participants formed the QT/QTc Set.
Arm/Group | Moxifloxacin (QT/QTc Set)
Number analyzed (Participants) | 47
milliseconds
  0.75 hour Predose | 0.9 [-1.2 to 3.0]
  0.5 hour Predose | 1.9 [-0.2 to 4.1]
  0.25 hour Predose | 2.4 [0.5 to 4.4]
  0.25 hour Postdose | 1.8 [-0.5 to 4.0]
  0.5 hour Postdose | 3.6 [1.4 to 5.8]
  1 hour Postdose | 8.6 [6.2 to 10.9]
  1.5 hours Postdose | 9.8 [7.3 to 12.2]
  2 hours Postdose | 10.6 [8.0 to 13.2]
  3 hours Postdose | 9.0 [5.8 to 12.3]
  4 hours Postdose | 9.0 [6.4 to 11.7]
  6 hours Postdose | 8.7 [6.3 to 11.2]
  8 hours Postdose | 8.6 [6.2 to 11.1]
  12 hours Postdose | 5.5 [2.3 to 8.7]
  18 hours Postdose | 7.9 [5.3 to 10.5]
  24 hours Postdose | 6.3 [3.8 to 8.7]

3. Secondary Outcome: Placebo-corrected Change From Baseline in Heart Rate (HR) Interval on Day 1
Description: Placebo-corrected change from Baseline in HR, (ΔΔHR) evaluated during the Target Dose Day of the padsevonil/moxifloxacin and placebo Treatment Periods, using linear mixed-effects model analysis.
Time Frame: Day 1 : 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: The QT/QTc Set included all study participants in the SS with measurements at Baseline as well as on-treatment with at least 1 postdose time point with a valid change-from Baseline QTcF (ΔQTcF) value. Here, number of participants were included who were evaluable for the assessment. The Target Dose for moxifloxacin was at Day 8. Therefore, the data was analyzed at Day 8 only.
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Padsevonil (QT/QTc Set) | Moxifloxacin (QT/QTc Set)
Number analyzed (Participants) | 50 | 0
beats per minute (bpm)
  Day 1: 0.25 hour Postdose | 0.2 [-0.8 to 1.2] |
  Day 1: 0.5 hour Postdose | 2.0 [0.6 to 3.4] |
  Day 1: 1 hour Postdose | 1.4 [0.0 to 2.8] |
  Day 1: 1.5 hours Postdose | -0.1 [-1.7 to 1.5] |
  Day 1: 2 hours Postdose | 0.1 [-1.6 to 1.9] |
  Day 1: 3 hours Postdose | -2.3 [-4.2 to -0.3] |
  Day 1: 4 hours Postdose | -2.0 [-3.9 to -0.1] |
  Day 1: 6 hours Postdose | 0.8 [-0.9 to 2.5] |
  Day 1: 8 hours Postdose | -2.0 [-3.7 to -0.3] |
  Day 1: 12 hours Postdose | 0.1 [-1.6 to 1.8] |
  Day 1: 24 hours Postdose | -0.8 [-2.2 to 0.6] |

4. Secondary Outcome: Placebo-corrected Change From Baseline in Heart Rate (HR) Interval on Day 8
Description: as for outcome 3
Time Frame: Day 8 : 0.75, 0.5, 0.25 predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Padsevonil (QT/QTc Set) | Moxifloxacin (QT/QTc Set)
Number analyzed (Participants) | 46 | 47
beats per minute (bpm)
  Day 8: 0.75 hour Predose | -2.0 [-3.7 to -0.2] | -0.4 [-1.9 to 1.2]
  Day 8: 0.5 hour Predose | -2.0 [-3.6 to -0.4] | 0.4 [-1.4 to 2.2]
  Day 8: 0.25 hour Predose | -1.1 [-2.9 to 0.6] | 0.5 [-1.3 to 2.3]
  Day 8: 0.25 hour Postdose | -1.1 [-2.8 to 0.6] | -0.4 [-1.6 to 0.8]
  Day 8: 0.5 hour Postdose | -2.0 [-3.7 to 0.4] | 0.1 [-1.5 to 1.6]
  Day 8: 1 hour Postdose | -1.9 [-3.5 to -0.3] | 1.9 [0.5 to 3.3]
  Day 8: 1.5 hours Postdose | -1.1 [-2.7 to 0.5] | 1.3 [-0.1 to 2.7]
  Day 8: 2 hours Postdose | -3.0 [-4.6 to -1.4] | 1.0 [-0.3 to 2.3]
  Day 8: 3 hours Postdose | -2.2 [-4.4 to 0.0] | -1.8 [-3.5 to -0.1]
  Day 8: 4 hours Postdose | -1.2 [-3.3 to 0.8] | -0.4 [-2.0 to 1.3]
  Day 8: 6 hours Postdose | -1.0 [-3.2 to 1.2] | 0.2 [-1.5 to 2.0]
  Day 8: 8 hours Postdose | -3.3 [-5.1 to -1.5] | 0.2 [-1.4 to 1.9]
  Day 8: 12 hours Postdose | -0.6 [-2.4 to 1.3] | 0.3 [-1.3 to 1.8]
  Day 8: 18 hours Postdose | 1.1 [-0.8 to 2.9] | 1.3 [-0.6 to 3.2]
  Day 8: 24 hours Postdose | -1.0 [-3.2 to 1.2] | 0.4 [-1.3 to 2.1]

5. Secondary Outcome: Placebo-corrected Change From Baseline for PR Interval on Day 1
Description: Placebo-corrected change from Baseline in PR, (ΔΔPR) evaluated during the Target Dose Day of the padsevonil/moxifloxacin and placebo Treatment Periods, using linear mixed-effects model analysis.
Time Frame: Day 1 : 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 3
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Padsevonil (QT/QTc Set) | Moxifloxacin (QT/QTc Set)
Number analyzed (Participants) | 50 | 0
milliseconds
  Day 1: 0.25 hour Postdose | -0.4 [-2.0 to 1.1] |
  Day 1: 0.5 hour Postdose | 0.5 [-1.2 to 2.3] |
  Day 1: 1 hour Postdose | 2.2 [0.2 to 4.2] |
  Day 1: 1.5 hours Postdose | 1.9 [-0.2 to 3.9] |
  Day 1: 2 hours Postdose | 1.9 [-0.4 to 4.2] |
  Day 1: 3 hours Postdose | 2.2 [-0.3 to 4.7] |
  Day 1: 4 hours Postdose | 2.6 [-0.2 to 5.4] |
  Day 1: 6 hours Postdose | 2.3 [-0.7 to 5.3] |
  Day 1: 8 hours Postdose | 3.5 [0.9 to 6.1] |
  Day 1: 12 hours Postdose | 1.3 [-1.8 to 4.3] |
  Day 1: 24 hours Postdose | 1.3 [-0.8 to 3.4] |

6. Secondary Outcome: Placebo-corrected Change From Baseline for PR Interval on Day 8
Description: as for outcome 5
Time Frame: Day 8 : 0.75, 0.5, 0.25 predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Padsevonil (QT/QTc Set) | Moxifloxacin (QT/QTc Set)
Number analyzed (Participants) | 46 | 47
milliseconds
  Day 8: 0.75 hour Predose | 2.4 [-0.4 to 5.2] | -0.6 [-3.5 to 2.3]
  Day 8: 0.5 hour Predose | 1.8 [-0.7 to 4.3] | -1.0 [-3.7 to 1.7]
  Day 8: 0.25 hour Predose | 1.2 [-1.5 to 4.0] | -1.2 [-4.1 to 1.7]
  Day 8: 0.25 hour Postdose | 2.4 [-0.4 to 5.2] | -0.4 [-3.1 to 2.4]
  Day 8: 0.5 hour Postdose | 3.1 [0.2 to 6.0] | -1.6 [-4.3 to 1.1]
  Day 8: 1 hour Postdose | 3.8 [1.1 to 6.6] | -0.8 [-3.3 to 1.7]
  Day 8: 1.5 hours Postdose | 4.2 [1.4 to 7.0] | -0.8 [-3.3 to 1.7]
  Day 8: 2 hours Postdose | 3.6 [1.0 to 6.3] | -1.3 [-3.7 to 1.2]
  Day 8: 3 hours Postdose | 3.6 [0.6 to 6.6] | -3.1 [-6.1 to 0.0]
  Day 8: 4 hours Postdose | 4.1 [1.1 to 7.2] | -3.3 [-6.2 to -0.3]
  Day 8: 6 hours Postdose | 3.3 [0.5 to 6.2] | -2.3 [-4.9 to 0.4]
  Day 8: 8 hours Postdose | 2.6 [-0.5 to 5.7] | -2.3 [-4.8 to 0.2]
  Day 8: 12 hours Postdose | 1.6 [-2.0 to 5.3] | -2.9 [-6.0 to 0.1]
  Day 8: 18 hours Postdose | -0.2 [-3.7 to 3.2] | -2.1 [-5.3 to 1.1]
  Day 8: 24 hours Postdose | -0.6 [-2.1 to 3.3] | -1.9 [-4.8 to 0.9]

7. Secondary Outcome: Placebo-corrected Change From Baseline for QRS Interval on Day 1
Description: Placebo-corrected change from Baseline for QRS interval, (ΔΔQRS) evaluated during the Target Dose Day of the padsevonil/moxifloxacin and placebo Treatment Periods, using linear mixed-effects model analysis.
Time Frame: Day 1 : 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose
Population: as for outcome 3
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Padsevonil (QT/QTc Set) | Moxifloxacin (QT/QTc Set)
Number analyzed (Participants) | 50 | 0
milliseconds
  Day 1: 0.25 hour Postdose | -0.2 [-0.4 to 0.1] |
  Day 1: 0.5 hour Postdose | -0.1 [-0.4 to 0.1] |
  Day 1: 1 hour Postdose | 0.0 [-0.2 to 0.3] |
  Day 1: 1.5 hours Postdose | -0.2 [-0.5 to 0.1] |
  Day 1: 2 hours Postdose | -0.3 [-0.6 to 0.1] |
  Day1: 3 hours Postdose | -0.3 [-0.7 to 0.0] |
  Day 1: 4 hours Postdose | -0.2 [-0.7 to 0.1] |
  Day1: 6 hours Postdose | -0.1 [-0.6 to 0.4] |
  Day1: 8 hours Postdose | -0.3 [-0.7 to 0.2] |
  Day1: 12 hours Postdose | 0.1 [-0.6 to 0.7] |
  Day1: 24 hours Postdose | -0.3 [-0.6 to 0.1] |

8. Secondary Outcome: Placebo-corrected Change From Baseline for QRS Interval on Day 8
Description: as for outcome 7
Time Frame: Day 8 : 0.75, 0.5, 0.25 predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Padsevonil (QT/QTc Set) | Moxifloxacin (QT/QTc Set)
Number analyzed (Participants) | 46 | 47
milliseconds
  Day 8: 0.75 hour Predose | -0.2 [-0.9 to 0.6] | 0.0 [-0.7 to 0.8]
  Day 8: 0.5 hour Predose | -0.1 [-0.9 to 0.6] | 0.0 [-0.7 to 0.7]
  Day 8: 0.25 hour Predose | -0.1 [-0.8 to 0.6] | 0.2 [-0.5 to 0.9]
  Day 8: 0.25 hour Postdose | -0.2 [-1.0 to 0.5] | -0.1 [-0.8 to 0.7]
  Day 8: 0.5 hour Postdose | -0.2 [-1.0 to 0.5] | -0.1 [-0.9 to 0.6]
  Day 8: 1 hour Postdose | -0.5 [-1.2 to 0.3] | 0.0 [-0.8 to 0.8]
  Day 8: 1.5 hours Postdose | -0.6 [-1.3 to 0.2] | -0.1 [-0.8 to 0.7]
  Day 8: 2 hours Postdose | -0.2 [-1.0 to 0.6] | 0.1 [-0.7 to 0.8]
  Day 8: 3 hours Postdose | -0.2 [-0.9 to 0.6] | 0.1 [-0.5 to 0.8]
  Day 8: 4 hours Postdose | -0.3 [-1.1 to 0.4] | 0.0 [-0.7 to 0.7]
  Day 8: 6 hours Postdose | -0.4 [-1.2 to 0.4] | -0.1 [-0.8 to 0.7]
  Day 8: 8 hours Postdose | 0.0 [-0.8 to 0.8] | 0.0 [-0.7 to 0.6]
  Day 8: 12 hours Postdose | -0.2 [-1.0 to 0.6] | 0.5 [-0.4 to 1.3]
  Day 8: 18 hours Postdose | -1.1 [-2.0 to -0.2] | -0.1 [-1.0 to 0.8]
  Day 8: 24 hours Postdose | -0.1 [-0.7 to 0.6] | 0.8 [0.1 to 1.5]

9. Secondary Outcome: Number of Participants With Treatment-emergent Changes for T-wave Morphology and U-wave Presence
Description: Number of Participants with treatment-emergent changes of electrocardiogram waveforms as T-waves and U-waves. If a given morphology occurs multiple times at a given time point, that occurrence was only counted 1 time for that time point. If more than 1 morphology type was observed at a given time point, both morphology types were counted. A subject can appear in more than 1 category.
Time Frame: Day 8 : 0.75, 0.5, 0.25 hours predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24 hours postdose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (QT/QTc Set): Participants received placebo matched to PSL Treatment Period doses, bid up to Day 11. Participants formed the QT/QTc Set.
Arm/Group | Padsevonil (QT/QTc Set) | Moxifloxacin (QT/QTc Set) | Placebo (QT/QTc Set)
Number analyzed (Participants) | 51 | 47 | 50
Participants
  Flat | 0 | 0 | 0
  Notched (+) | 0 | 0 | 0
  Biphasic | 1 | 0 | 0
  Normal (-) | 0 | 0 | 0
  Notched (-) | 0 | 0 | 0
  U-Wave Presence | 0 | 1 | 1

10. Secondary Outcome: Change From Baseline in QTcF Evaluated at Drug-specific Tmax for Padsevonil
Description: Change from Baseline in QTcF (ΔQTcF) evaluated at drug-specific tmax (Δtmax) for padsevonil, using an analysis of variance (ANOVA) mixed-effect model.
Time Frame: Day 8 : 0.75, 0.5, 0.25 hours predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18 hours postdose
Population: The QT/QTc Set included all study participants in the SS with measurements at Baseline as well as on-treatment with at least 1 postdose time point with a valid change-from Baseline QTcF (ΔQTcF) value.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Arm/Group | Padsevonil (QT/QTc Set)
Number analyzed (Participants) | 51
milliseconds | -1.0 [-3.7 to 1.6]

11. Secondary Outcome: Change From Baseline in QTcF Evaluated at Drug-specific Tmax for Metabolite 1
Description: Change from Baseline in QTcF (ΔQTcF) evaluated at drug-specific tmax (Δtmax) for metabolite 1, using an analysis of variance (ANOVA) mixed-effect model.
Time Frame: Day 8 : 0.75, 0.5, 0.25 hours predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18 hours postdose
Population: as for outcome 10
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- Metabolite 1 (QT/QTc Set): Participants received PSL (padsevonil metabolite 1) 100 mg to 400 mg orally bid during the 11 Days PSL Treatment Period. On Day 8, the Target Dose Day, participants received PSL 400 mg in the morning only and placebo in the afternoon. Participants formed the QT/QTc Set.
Arm/Group | Metabolite 1 (QT/QTc Set)
Number analyzed (Participants) | 51
milliseconds | 0.1 [-2.3 to 2.5]

12. Secondary Outcome: Change From Baseline in QTcF Evaluated at Drug-Specific Tmax for Metabolite 2
Description: Change from Baseline in QTcF (ΔQTcF) evaluated at drug-specific tmax (Δtmax) for metabolite 2, using an analysis of variance (ANOVA) mixed-effect model.
Time Frame: Day 8 : 0.75, 0.5, 0.25 hours predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18 hours postdose
Population: as for outcome 10
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds
Groups:
- Metabolite 2 (QT/QTc Set): Participants received PSL (padsevonil metabolite 2) 100 mg to 400 mg orally bid during the 11 Days PSL Treatment Period. On Day 8, the Target Dose Day, participants received PSL 400 mg in the morning only and placebo in the afternoon. Participants formed the QT/QTc Set.
Arm/Group | Metabolite 2 (QT/QTc Set)
Number analyzed (Participants) | 51
milliseconds | -1.0 [-3.5 to 1.5]

13. Secondary Outcome: Maximum Observed Plasma Concentration at Steady State (Cmax, ss) for Padsevonil
Description: Cmax,ss: Maximum observed plasma concentration of padsevonil at steady state.
Time Frame: Day 8: 0.5 hours predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18 hours postdose
Population: The PKS included all study participants who received at least 1 dose of study medication, had no important Protocol deviations affecting the PK, and for whom at least 1 measurable PK concentration was available. Here, number of participants were included who were evaluable for the assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram per milliliter (ng/ml)
Groups:
- Padsevonil (PKS): Participants received PSL 100 mg to 400 mg orally bid during the 11 Days PSL Treatment Period.
  On Day 8, the Target Dose Day, participants received PSL 400 mg in the morning only and placebo in the afternoon. Participants formed Pharmacokinetic Set (PKS).
Arm/Group | Padsevonil (PKS)
Number analyzed (Participants) | 47
nanogram per milliliter (ng/ml) | 2119 [1912 to 2348]

14. Secondary Outcome: Time of Observed Maximum Concentration (Tmax) at Steady State for Padsevonil
Description: tmax: Time of observed maximum plasma concentration at steady state.
Time Frame: Day 8: 0.5 hours predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18 hours postdose
Population: as for outcome 13
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Padsevonil (PKS)
Number analyzed (Participants) | 47
hours (h) | 0.5100 [0.250 to 4.00]

15. Secondary Outcome: Area Under the Plasma Concentration Time Curve (AUCtau) at Steady State for Padsevonil
Description: AUCtau: Area under the plasma concentration time curve over a dosing interval at steady state.
Time Frame: Day 8: 0.5 hours predose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18 hours postdose
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Padsevonil (PKS)
Number analyzed (Participants) | 47
hour*nanogram per milliliter (h*ng/mL) | 8586 [7752 to 9510]

16. Secondary Outcome: Percentage of Participants With Adverse Events From Baseline to Safety Follow-up (up to Day 67)
Description: An Adverse Event is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage.
Time Frame: From Baseline to Safety Follow-up (up to Day 67)
Population: Safety Set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Groups:
- Padsevonil (SS): Participants received PSL 100 mg to 400 mg orally bid during the 11 Days PSL Treatment Period. On Day 8, the Target Dose Day, participants received PSL 400 mg in the morning only and placebo in the afternoon. Participants formed Safety Set (SS).
- Moxifloxacin (SS): Participants received placebo matched to PSL Treatment Period doses, bid up to Day 11. On Day 8, the Target Dose Day, participants received MXF 400 mg in the morning and placebo in the afternoon. Participants formed the SS.
- Placebo (SS): Participants received placebo matched to PSL Treatment Period doses, bid up to Day 11. Participants formed the SS.
Arm/Group | Padsevonil (SS) | Moxifloxacin (SS) | Placebo (SS)
Number analyzed (Participants) | 51 | 51 | 50
percentage of participants | 88.2 | 31.4 | 20.0

17. Secondary Outcome: Percentage of Participants With Serious Adverse Events From Baseline to Safety Follow-up (up to Day 67)
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline to Safety Follow-up (up to Day 67)
Population: Safety Set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Padsevonil (SS) | Moxifloxacin (SS) | Placebo (SS)
Number analyzed (Participants) | 51 | 51 | 50
percentage of participants | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants With Treatment Related Adverse Events From Baseline to Safety Follow-up (up to Day 67)
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Baseline to Safety Follow-up (up to Day 67)
Population: Safety Set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Padsevonil (SS) | Moxifloxacin (SS) | Placebo (SS)
Number analyzed (Participants) | 51 | 51 | 50
percentage of participants | 86.3 | 5.9 | 4.0

19. Secondary Outcome: Percentage of Participants With Adverse Events Leading to Discontinuation of the Study From Baseline to Safety Follow-up (up to Day 67)
Description: An Adverse Event is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage. The results of this Primary Outcome Measure are summarized from the Adverse Event pages of the Case Report Forms.
Time Frame: From Baseline to Safety Follow-up (up to Day 67)
Population: Safety Set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Padsevonil (SS) | Moxifloxacin (SS) | Placebo (SS)
Number analyzed (Participants) | 51 | 51 | 50
percentage of participants | 2.0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline to Safety Follow Up (up to Day 67)
Description: Any AE that starts on or after the date of the first dose of study drug and on or before the last date of the last treatment period or any unresolved event already present before administration of treatment that worsens in intensity following exposure to the treatment.
Arm/Group | Padsevonil (SS) | Moxifloxacin (SS) | Placebo (SS)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 38/51 | 13/51 | 7/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Padsevonil (SS) (N=51) | Moxifloxacin (SS) (N=51) | Placebo (SS) (N=50)
Diplopia (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Medical device site reaction (General disorders) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 21 (22) | 2 (2) | 0 (0)
Sedation (Nervous system disorders) | 15 (15) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 9 (13) | 5 (6) | 5 (5)
Somnolence (Nervous system disorders) | 8 (8) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 4 (4) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT04126343/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT04126343/SAP_001.pdf